CLINICAL TRIAL: NCT05920707
Title: Common and Differentiated Representations Between Social Exclusion and Social Separation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Weihua Zhao, Associate Professor, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: UESTC-neuSCAN-93
Record Dates: First submitted 2023-06-02; First posted 2023-06-27 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Healthy
Keywords: Social exclusion; Social separation; Oxytocin; Arginine Vasopressin; fMRI
MeSH Terms: conditions — Social Isolation; Diabetes Insipidus

STUDY DESIGN:
Intervention Model Description: Randomized placebo-controlled double-blind between-subject design
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intranasal Oxytocin (Active Comparator): Administer oxytocin (24 IU) intranasally.
  Interventions: Drug: Intranasal Oxytocin
- Intranasal Arginine Vasopressin (Active Comparator): Administer Arginine Vasopressin (20 IU) intranasally.
  Interventions: Drug: Intranasal Arginine Vasopressin
- Intranasal placebo (Placebo Comparator): Administer placebo intranasally.
  Interventions: Drug: Intranasal placebo
- Intranasal nothing (control) (No Intervention): Control condition

INTERVENTIONS:
Drug: Intranasal Oxytocin — Administer oxytocin (24 IU) intranasally, 6 individual 0.1 ml puffs (4 IU/0. 1ml), three puffs per nostril one every 30 seconds.
  Arms: Intranasal Oxytocin
Drug: Intranasal Arginine Vasopressin — Administer arginine vasopressin (20 IU) intranasally, 6 individual 0.1 ml puffs (3.33 IU/0. 1ml), three puffs per nostril one every 30 seconds.
  Arms: Intranasal Arginine Vasopressin
Drug: Intranasal placebo — Administer placebo intranasally, 6 individual 0.1 ml puffs, three puffs per nostril one every 30 seconds.
  Arms: Intranasal placebo

SUMMARY:
Explore the shared or separated neural mechanisms of social exclusion and social segregation and compare differential effects of AVP and OXT on these social interaction function.

DETAILED DESCRIPTION:
A large body of research has shown that there are differences in the neural representation between social exclusion and social segregation, but the results are inconsistent, and the exploration of the neural basis is still insufficient. In addition, there are two mainstream theoretical explanations for these differences, namely the construction-level theory and the emotion-based theory, but there is no consistent theoretical model yet. Therefore, further exploration is necessary to confirm the cognitive and neural mechanisms underlying the differences between social exclusion and social segregation, and to attempt to reveal the theoretical explanations for these differences. In this project, the investigators propose to perform behavioral and functional magnetic resonance imaging (fMRI) techniques to examine the shared or separate neural mechanisms of social exclusion and social segregation (exp 1: social exclusion; exp 2: social separation) and investigate the modulatory effects of OXT/AVP on them (PLC/24IU OXT/20IU AVP).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects;
2. Without any past or present psychiatric or neurological disorders;
3. Without any current psychotherapeutic medication.

EXclusion Criteria:

1. With any past or present psychiatric or neurological disorders;
2. With any current psychotherapeutic medication.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-04-20 (Actual); Primary Completion 2023-09-20 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Neural index: OXT and AVP effects on fMRI based- social exclusion and social separation tasks | 45 minutes after treatment administration
  Comparions between OXT and AVP on social exclusion and social separation on brain activity or representations
Behavioral index: behavioral ratings of social exclusion and social separation tasks | Immediately after fMRI scanning
  Comparions between social exclusion and social separation in pain ratings

CONTACTS AND LOCATIONS:
Overall Officials: Siying Wang, Dr, Study Chair — University of Electronic Science and Technology of China
Locations (1):
- University of Electronic Science and Technology of China(UESTC), Chengdu, Sichuan, China